CLINICAL TRIAL: NCT06345235
Title: Assessment of the Association of New Biomarkers (GDF15, ST2, Galectin-3, TIMP-1, MMP-9, NfL) and Plasma Prothrombotic Potential in the Course of Cardiac Transthyretin Amyloidosis
Brief Title: New Biomarkers and Plasma Prothrombotic Potential in Cardiac Transthyretin Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Other Study IDs: ID DEC-2023/07/X/NZ5/00141
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Transthyretin Amyloidosis
Keywords: transthyretin amyloidosis; GDF15; ST2; galectin-3; TIMP-1; MMP-9; NfL; plasma prothrombotic potential; amyloidosis; cardiomyopathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis; Cardiomyopathies | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- with ATTR cardiomyopthy: blood sample
  Interventions: Diagnostic Test: blood test
- TTR variant carier and no ATTR cardiomyopthy: blood sample
  Interventions: Diagnostic Test: blood test
- controls: blood sample
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — Assessment of the association of new biomarkers (GDF15, ST2, galectin-3, TIMP-1, MMP-9, NfL) and plasma prothrombotic potential in groups 1, 2, 3

SUMMARY:
The development of cardiac amyloidosis is caused by the deposition of misfolded, insoluble proteins in the extracellular matrix of tissues. An important element of the clinical picture of the disease is the increased risk of thromboembolic complications, independent of the occurrence of atrial fibrillation, and the presence of intracardiac thrombi. The pathomechanism may be related to an increase in filling pressure or amyloid infiltration leading to myocardial damage and endothelial dysfunction, which may activate the prothrombotic inflammatory cascade, resulting in increased thrombogenic potential. Currently, there is limited published data on the potential role of new heart failure biomarkers in the assessment of ATTR cardiomyopathy, particularly in the assessment of asymptomatic carriers of pathogenic TTR variants. Moreover, there are few literature reports on the direct assessment of the coagulation system in this group of patients, and the pathomechanism of the increased thromboembolic risk is unexplored.

Purpose of the study: To assess the diagnostic value of biomarkers related to heart failure (growth differentiation factor-15 (GDF15), soluble suppression of tumorigenicity-2 (ST2), galectin-3), amyloidosis ( TTR, tissue inhibitor of metalloproteinase-1 (TIMP-1), matrix metalloproteinase-9 (MMP-9, matrix metalloproteinase-9), neurofilament light chain (NfL)) and the generation potential thrombin as a marker of the prothrombotic state in the course of ATTR.

Methods: This prospective, single-center study will include consecutive patients diagnosed with ATTR cardiomyopathy (GROUP 1, n=30), asymptomatic carriers of pathogenic TTR variants (GROUP 2, n=30), and a matched control group of healthy volunteers (GROUP 3 , n=20). Material for research was collected and secured from all study participants. After giving informed consent, all patients will be tested using the ELISA method from peripheral blood (enzyme-linked immunosorbent assay) GDF15, ST2, TTR, TIMP-1, MMP-9, galectin-3, NfL. The values of these biomarkers will be compared in subgroups and correlated with clinical data, laboratory test results, echocardiography including analysis of left ventricular global strain (GLS), and scintigraphy. Additionally, the prothrombotic potential of plasma will be tested in both groups of patients using the calibrated automatic thrombogram (CAT) method, in accordance with the protocol previously used in the laboratory Expected results: The project will provide information on the value of biomarkers in the assessment of ATTR cardiomyopathy, especially in the assessment of asymptomatic carriers of pathogenic TTR variants, which may translate into the creation of a diagnostic algorithm for early identification of the development of the disease. Moreover, it will allow us to determine whether patients with cardiac ATTR are characterized by a prothrombotic state, which has not yet been described in the literature and may have potential clinical implications.

DETAILED DESCRIPTION:
Introduction: The development of cardiac amyloidosis is caused by the deposition of misfolded, insoluble proteins in the extracellular matrix of tissues. More than 30 precursor proteins can form amyloid fibrils, but two types account for 95% of cases of amyloid cardiomyopathy (CA): immunoglobulin light chain (AL) amyloidosis and transthyretin amyloidosis (ATTR). There are two forms of ATTR - acquired wild-type ATTR (ATTRwt) and the hereditary form (ATTRm), developing on the basis of mutations in the transthyretin (TTR) gene. Among patients with CA, as the disease progresses, heart failure develops, and if left untreated, the disease leads to death within 6 months to 3 years. Due to the unique pathology of the disease, the clinical picture includes the development of: peripheral polyneuropathy, autonomic dysfunction, and an increased risk of thromboembolic complications. An important element of the clinical picture of the disease is the increased risk of thromboembolic complications, independent of the occurrence of atrial fibrillation, and the presence of intracardiac thrombi. The pathomechanism may be related to an increase in filling pressure or amyloid infiltration leading to myocardial damage and endothelial dysfunction, which may activate the prothrombotic inflammatory cascade, resulting in increased thrombogenic potential. Scintigraphy has become a key technique in identifying patients with ATTR - in the absence of a detectable monoclonal protein, it allows for a non-invasive diagnosis of ATTR. Due to the development of disease-specific therapies (stabilizing drugs, gene therapy), it is important to diagnose the disease at an early stage, when the symptoms are relatively mild, and the implementation of treatment allows to stop the development of the disease and reduce mortality. Currently, there is limited published data on the potential role of new heart failure biomarkers in the assessment of ATTR cardiomyopathy, particularly in the assessment of asymptomatic carriers of pathogenic TTR variants. Moreover, there are few literature reports on the direct assessment of the coagulation system in this group of patients, and the pathomechanism of the increased thromboembolic risk is unexplored.

Purpose of the study: To assess the diagnostic value of biomarkers related to heart failure (growth differentiation factor-15 (GDF15), soluble suppression of tumorigenicity-2 (ST2), galectin-3), amyloidosis (TTR, tissue inhibitor of metalloproteinase-1 (TIMP-1), matrix metalloproteinase-9 (MMP-9, matrix metalloproteinase-9), neurofilament light chain (NfL)) and the generation potential thrombin as a marker of the prothrombotic state in the course of ATTR.

Methods: This prospective, single-center study will include consecutive patients diagnosed with ATTR cardiomyopathy (GROUP 1, n=30), asymptomatic carriers of pathogenic TTR variants (GROUP 2, n=30), and a matched control group of healthy volunteers (GROUP 3 , n=20). Material for research was collected and secured from all study participants. After giving informed consent, all patients will be tested using the ELISA method from peripheral blood (enzyme-linked immunosorbent assay) GDF15, ST2, TTR, TIMP-1, MMP-9, galectin-3, NfL. The values of these biomarkers will be compared in subgroups and correlated with clinical data, laboratory test results, echocardiography including analysis of left ventricular global strain (GLS), and scintigraphy. Additionally, the prothrombotic potential of plasma will be tested in both groups of patients using the calibrated automatic thrombogram (CAT) method, in accordance with the protocol previously used in the laboratory. The results will be compared with reference values for the control group. All tests will be performed by qualified and experienced staff.

Expected results: The project will provide information on the value of biomarkers in the assessment of ATTR cardiomyopathy, especially in the assessment of asymptomatic carriers of pathogenic TTR variants, which may translate into the creation of a diagnostic algorithm for early identification of the development of the disease. Moreover, it will allow us to determine whether patients with cardiac ATTR are characterized by a prothrombotic state, which has not yet been described in the literature and may have potential clinical implications. The obtained results can be used as starting data for further research on the coagulation system in ATTR in subsequent scientific projects.

ELIGIBILITY:
Inclusion Criteria:

the study will include consecutive patients diagnosed with ATTR cardiomyopathy (GROUP 1, n=30), asymptomatic carriers of pathogenic TTR variants (GROUP 2, n=30), and a matched control group of healthy volunteers (GROUP 3, n=20)

1. age over 18
2. expressing informed written consent
3. clinical criteria (one of the following for a given group):

   1. ATTR cardiomyopathy (GROUP 1),
   2. asymptomatic carrier of the pathogenic variant of the TTR gene (GROUP 2),
   3. no diagnosed ATTR cardiomyopathy and no pathogenic variant of the TTR gene (GROUP 3).

Exclusion criteria:

1. age under 18 years of age
2. failure to provide informed written consent
3. pregnancy and lactation

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 consecutive patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-07-11 (Estimated); Study Completion 2024-07-11 (Estimated)

PRIMARY OUTCOMES:
Biomarkers | baseline evaluation at the day of enrolment
  To assess the diagnostic value of growth differentiation factor-15 (GDF15) in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.
Thrombin as a marker | baseline evaluation at the day of enrolment
  To assess the generation potential thrombin as a marker of the prothrombotic state in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group
Biomarkers | baseline evaluation at the day of enrolment
  To assess the diagnostic value of soluble suppression of tumorigenicity-2 (ST2) in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.
Biomarkers | baseline evaluation at the day of enrolment
  To assess the diagnostic value of galectin-3 in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.
Biomarkers | baseline evaluation at the day of enrolment
  To assess the diagnostic value of tissue inhibitor of metalloproteinase-1 (TIMP-1) in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.
Biomarkers | baseline evaluation at the day of enrolment
  To assess the value of TTR in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.
Biomarkers | baseline evaluation at the day of enrolment
  To assess the diagnostic value of matrix metalloproteinase-9 (MMP-9)in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.
Biomarkers | baseline evaluation at the day of enrolment
  To assess the diagnostic value of neurofilament light chain (NfL) in the course of ATTR compared to asymptomatic pathogenic TTR variant gene carriers and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- John Paul II Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawor M, Holcman K, Franaszczyk M, Lipowska M, Michalek P, Teresinska A, Bilinska ZT, Rubis P, Kostkiewicz M, Szot W, Podolec P, Grzybowski J. Spectrum of transthyretin gene mutations and clinical characteristics of Polish patients with cardiac transthyretin amyloidosis. Cardiol J. 2022;29(6):985-993. doi: 10.5603/CJ.a2020.0104. Epub 2020 Aug 13. PMID 32789836
- [Background] Holcman K, Dziuk M, Grzybowski J, Teresinska A, Malkowski B, Jedrzejuk D, Brockhuis B, Czepczynski R, Tomkiewicz-Pajak L, Kostkiewicz M. The scintigraphic diagnosis of cardiac amyloidosis. An expert opinion endorsed by the Section of Nuclear Medicine of the Polish Cardiac Society and the Polish Nuclear Medicine Society. Nucl Med Rev Cent East Eur. 2022;25(2):142-147. doi: 10.5603/NMR.a2022.0033. PMID 35929128
- [Background] Ticau S, Sridharan GV, Tsour S, Cantley WL, Chan A, Gilbert JA, Erbe D, Aldinc E, Reilly MM, Adams D, Polydefkis M, Fitzgerald K, Vaishnaw A, Nioi P. Neurofilament Light Chain as a Biomarker of Hereditary Transthyretin-Mediated Amyloidosis. Neurology. 2021 Jan 19;96(3):e412-e422. doi: 10.1212/WNL.0000000000011090. Epub 2020 Oct 21. PMID 33087494
- [Background] Castiglione V, Franzini M, Aimo A, Carecci A, Lombardi CM, Passino C, Rapezzi C, Emdin M, Vergaro G. Use of biomarkers to diagnose and manage cardiac amyloidosis. Eur J Heart Fail. 2021 Feb;23(2):217-230. doi: 10.1002/ejhf.2113. Epub 2021 Feb 21. PMID 33527656
- [Background] Garcia-Pavia P, Rapezzi C, Adler Y, Arad M, Basso C, Brucato A, Burazor I, Caforio ALP, Damy T, Eriksson U, Fontana M, Gillmore JD, Gonzalez-Lopez E, Grogan M, Heymans S, Imazio M, Kindermann I, Kristen AV, Maurer MS, Merlini G, Pantazis A, Pankuweit S, Rigopoulos AG, Linhart A. Diagnosis and treatment of cardiac amyloidosis: a position statement of the ESC Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2021 Apr 21;42(16):1554-1568. doi: 10.1093/eurheartj/ehab072. PMID 33825853
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827